CLINICAL TRIAL: NCT01895179
Title: Time-Restricted Feeding to Improve Glucose Tolerance and Vascular Condition
Brief Title: Comparison of Time-Restricted Feeding Versus Grazing
Acronym: TIMED EATING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Courtney Peterson, Instructor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PBRC 13017
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Prediabetes; Insulin Resistance; Vascular Diseases
Keywords: Time-restricted feeding; Intermittent fasting; Prediabetes; Insulin resistance; Glucose tolerance; Insulin sensitivity; Circadian rhythms; Diurnal
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Vascular Diseases; Intermittent Fasting

ARMS (2):
- Time-Restricted Feeding (early in the day eating) (Experimental): Participants will consume all meals early in the day and within a 6-hour window.
  Interventions: Other: Time-Restricted Feeding
- Grazing (Placebo Comparator): Participants will eat meals spread out over the course of the day.
  Interventions: Other: Grazing

INTERVENTIONS:
Other: Time-Restricted Feeding — Time-restricted feeding is a variant of intermittent fasting that involves eating all of one's calories within a few hours each day (typically 4-9 hours), followed by a daily fast of 15-20 hours.
  Arms: Time-Restricted Feeding (early in the day eating)
Other: Grazing — Grazing involves eating meals spread out over the course of the day.
  Arms: Grazing

SUMMARY:
The purpose of this pilot study is to find out what eating meals in a short time period early in the day (time-restricted feeding) versus eating meals spread out during the day (grazing) does to the body's ability to control blood sugar and to the health of its blood vessels.

The investigators hypothesize that time-restricted feeding will be more effective at improving glucose tolerance and vascular condition (inflammation and micro- and macro-vascular function) than grazing.

DETAILED DESCRIPTION:
Each participant will eat according to one of the two eating schedules (grazing or time-restricted feeding) for 5 weeks, have a 7-week washout period, and then eat according to the other eating schedule for 5 weeks. Measurements of glucose homeostasis and vascular condition will be performed before and after a participant follows each eating schedule.

ELIGIBILITY:
Inclusion Criteria:

* Are male
* Overweight: Have a body mass index between 25 and 50 kg/m^2 inclusive (a number calculated from height and weight)
* Are 35-70 years of age
* Have a hemoglobin A1C between 5.5 - 6.4% or prior medical indication of prediabetes
* Have a blood sugar level between 140 and 199 mg/dL two hours after drinking a sugary solution (OGTT)
* Have been eating dinner at least 8.5 hours after eating breakfast at least 90% of the time during the past year
* Have not fasted (go for a day without any food) more than 12 days total during the past year
* Be willing to eat most meals at Pennington Biomedical and/or under supervision
* Not eat any food other than that served by Pennington Biomedical
* Not drink any alcohol, juice, or other beverages that have calories other than what is served by Pennington Biomedical
* Keep water and no-calorie drinks like tea or diet soda the same during both of the timed eating periods
* Be willing to eat your meals according to the fixed schedules

Exclusion Criteria:

* Have diabetes or are on anti-diabetes medication
* Have evidence of cardiovascular disease
* Suffer from significant cardiovascular, renal (kidney), cardiac (heart), liver, lung or nervous system disease
* Evidence of significant gastrointestinal issues or surgery that impacts nutrient absorption
* Regularly use medications such as steroids, beta blockers, and adrenergic-stimulating agents
* Are on any regular medicine that has not had the same dose for 1 month or longer
* Have a clinically significant abnormality as measured by a blood test
* Regularly drink alcohol (more than 2 servings per day)
* Have to do any kind of heavy physical activity
* Currently perform overnight shift work more than one day a week
* Are not able to eat only the food served to you by Pennington Biomedical, while in the study
* Are not able to stop drinking alcohol or other drinks with calories (e.g., soda, juice) other than what is served to you by Pennington Biomedical, while in the study

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-07; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in Glucose Tolerance | Before and after 5 weeks on each feeding schedule
  Glucose tolerance and indices of glucose homeostasis will be determined using an Oral Glucose Tolerance Test (OGTT).

SECONDARY OUTCOMES:
Change in Vascular Function | Before and after 5 weeks on each feeding schedule
  Macro- and micro-vascular function will be assessed by Radial Artery Applanation Tonometry and by Orthogonal Polarization Spectroscopy. The endpoints measured by these two tests include aortic blood pressure, arterial stiffness, capillary density, and red blood cell velocity.
Change in Inflammation and Metabolic Markers | Before and after 5 weeks on each feeding schedule
  Serum markers of inflammation, such as C-Reactive Protein (CRP) and inflammatory cytokines, and of metabolic processes will be measured (composite measure).

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717